CLINICAL TRIAL: NCT04666155
Title: A Randomised Controlled Trial to Evaluate Effectiveness and Cost-Effectiveness of Intermittent Colonic Exoperistalsis Treatment With MOWOOT Medical Device in Adults With Chronic Constipation Using Trans-Anal Irrigation.
Brief Title: MOWOOT Device Treatment for Adults With Chronic Constipation
Acronym: MOTACC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: usMIMA S.L. (Industry)
Collaborators: County Durham and Darlington NHS Foundation Trust (Other Government); University of York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MOW-06-2023
Record Dates: First submitted 2020-12-07; First posted 2020-12-14 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Constipation - Functional; Constipation-predominant Irritable Bowel Syndrome; Constipation Chronic Idiopathic; Constipation; Neurogenic; Constipation
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intermittent Colon Exoperistalsis (ICE) (Experimental): Intermittent Colon Exoperistalsis (ICE) Treatment with Mowoot device. 20min daily for 12 weeks
  Interventions: Device: Intermittent Colonic Exoperistalsis with MOWOOT device; Device: Standard of care with Trans-Anal Irrigation
- Standard-of-care with Trans-anal Irrigation (Soc TAI) (Active Comparator): Standard-of-care with Trans-anal Irrigation (Soc TAI) for chronic constipation for 12 weeks.
  Interventions: Device: Standard of care with Trans-Anal Irrigation

INTERVENTIONS:
Device: Intermittent Colonic Exoperistalsis with MOWOOT device — Patients under the experimental arm of the study should place the belt of the Mowoot device on the abdomen and use it for 20 minutes every day for 12 weeks. They should continue with their individualized standard of care againts constipation for the first 4 weeks. During the following 8 weeks of the interventional period of 12weeks, their use of SocTAI will be considered "rescue intervention". The 8weeks following the 12weeks of intervention, they can keep on using ICE device.or SocTAI or both.
  Arms: Intermittent Colon Exoperistalsis (ICE)
Device: Standard of care with Trans-Anal Irrigation — Patients under the active comparator arm of the study should continue with their individualized standard of care againts constipation for the 12weeks of intervention. The following 8 weeks they can keep on using SocTAI or ICE device or both.

SUMMARY:
The primary objective is to compare the effectiveness of the experimental Intermittent Colonic Exoperistalsis (ICE) treatment with MOWOOT, with the active control of trans-anal irrigation (TAI) as standard-of-care. The secondary objectives are to further compare the ICE treatment with MOWOOT to the TAI standard-of-care clinically and economically.

DETAILED DESCRIPTION:
The RCT will assess clinical effectiveness by means of quantitative and qualitative variables, and the cost effectiveness by means of economic outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Any gender 18 years or older
2. Symptoms meeting the American College of Gastroenterology definition of chronic constipation: unsatisfactory defaecation characterized by infrequent stool, difficult stool passage or both for at least previous 3 months
3. Bothered by their constipation
4. PAC-QOL ≥1.8
5. Using TAI for at least 3 months
6. Able to undertake the treatment with TAI or with the device themselves or with a carer willing to do it
7. Able to understand the study requirements
8. Able to understand written and spoken English (due to questionnaire validity)
9. Able and willing to provide written informed consent to participate

Exclusion Criteria:

Disease phenotype exclusion criteria:

1. Irritable Bowel Syndrome with Diarrhoea (IBS-D) or alternating constipation and diarrhoea (IBSmix): (not due to laxative use)
2. Inflammatory Bowel Disease (IBD)

   Device-related exclusion criteria:
3. Abdominal perimeter ≤65cm or ≥130cm
4. Unable to independently use the MOWOOT or TAI technology, unless a carer is available daily to assist

   Other medical conditions, medications and contraindications:
5. Previous large bowel resection
6. The presence of a stoma
7. External rectal prolapse
8. Active anorexia or bulimia
9. Active abdominal cancer
10. Large inguinal or umbilical hernia
11. Recent abdominal scars, abdominal wounds or skin disorders that may make abdominal massage uncomfortable
12. Pregnancy or attempt to become pregnant in the next 6 months
13. Use of strong opioids*
14. Use of antidepressants, bladder stabilisers or any other medication inducing, or treating, constipation unless used at a stable dose for at least 4 weeks before Screening Visit (this excludes laxatives which may be used as required up to three days before the screening visit)
15. Subjects already undertaking or have undertaken abdominal massage unless they underwent a previous washout period of at least 2 months
16. Participation in another parallel interventional clinical trial or less than 2 months from participation in a previous interventional clinical trial
17. Planned surgery for constipation if it might be within trial dates

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2024-04-25 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Changes in quality of life (PAC-QoL) | End of treatment (week 14, last week of treatment) - Baseline (before treatment)
  Semi-quantitative assessment of the changes in quality of life respect to chronic constipation, of patients using the ICE treatment with MOWOOT compared with patients under standard of care treatment. The measure is done according to PAC-QoL questionnaire.

SECONDARY OUTCOMES:
Frequency of use of TAI | Diary collected during the 2-week baseline period and for the last 2 weeks of the RCT period, and post-RCT period.
  How many days per week the patient has used TAI
Frequency of use of ICE | Diary collected during the 2-week baseline period and for the last 2 weeks of the RCT period, and post-RCT period.
  How many days per week the patient has used ICE
Changes in Constipation symptoms (PAC-SYM) | 3 times during the follow-up: Once at visit 1 (day 14 after recruitment), once at visit 2 (day 42 after treatment), and once more at visit 3 (day 154 after recruitment)
  Semi-quantitative assessment of the changes in symptoms of constipation of patients using the ICE treatment with MOWOOT compared with patients under standard of care treatment. The measure is done according to PAC-SYM questionnaire.
Changes in quality of life according to Euroqol ED5D5L | 3 times during the follow-up: Once at visit 1 (day 14 after recruitment), once at visit 2 (day 42 after treatment), and once more at visit 3 (day 154 after recruitment)
  Semi-quantitative assessment of the changes in self-perceived quality of life according to the EQ-5D-5L instrument
Changes in the number of days evacuation felt complete | Diary collected during the 2-week baseline period and for the last 2 weeks of the RCT period, and post-RCT period.
  Quantitative assessment of the change in the number of days per week evacuation felt complete at the end of the day
Changes in the maximum number of consecutive days without complete bowel movements | Diary collected during the 2-week baseline period and for the last 2 weeks of the RCT period, and post-RCT period.
  Quantitative assessment of the change in the maximum number of consecutive days within the 2-week diary period without complete bowel movementscomplete at the end of the day
Changes in the number of days with a normal stool | Diary collected during the 2-week baseline period and for the last 2 weeks of the RCT period, and post-RCT period.
  Quantitative assessment of the change in the number of days with a normal stool (Bristol Stool Scale 3-5) during the 2-week diary period
Changes in the mean time spent in bowel management | Diary collected during the 2-week baseline period and for the last 2 weeks of the RCT period, and post-RCT period.
  Quantitative assessment of the change in the mean time spent in bowel management per week
Changes in the mean time spent per evacuation | Diary collected during the 2-week baseline period and for the last 2 weeks of the RCT period, and post-RCT period.
  Quantitative assessment of the change in the mean time spent per evaquation
Changes in the number of days with fecal incontinence | Diary collected during the 2-week baseline period and for the last 2 weeks of the RCT period, and post-RCT period.
  Quantitative assessment of the change in the number of days with fecal incontinence per week
Changes in laxative use | Diary collected during the 2-week baseline period and for the last 2 weeks of the RCT period, and post-RCT period.
  Quantitative assessment of the change in the number of days per week taking laxatives
Changes in the use of SoC TAI (HE outcome) | Diary collected during the 2-week baseline period and for the last 2 weeks of the RCT period, and post-RCT period.
  Quantitative assessment of the changes in number of people (%) who stop using TAI while using ICE with MOWOOT during the 12-week RCT period; and mean/median change in the use of TAI while using Mowoot during the 12-week RCT period
Number of visits to GP and specialists (HE outcome) | 3 times during the follow-up: Once at visit 1 (day 14 after recruitment), once at visit 2 (day 42 after treatment), and once more at visit 3 (day 154 after recruitment)
  Quantitative assessment of the changes in the direct medical healthcare costs due to constipation-related problems assessed as the number of visits to GP and specialists (in primary care centres, hospitals, or visits received at home) over the previous 8 weeks
Number of visits to Accident & Emergency room (HE outcome) | 3 times during the follow-up: Once at visit 1 (day 14 after recruitment), once at visit 2 (day 42 after treatment), and once more at visit 3 (day 154 after recruitment)
  Quantitative assessment of the changes in the direct medical healthcare costs due to constipation-related problems assessed as the number of visits to to Accident & Emergency room (A&E) over the previous 8 weeks
  * Number of visits to GP and specialists (in primary care centres, hospitals, or visits received at home)
  * Number of visits to Accident & Emergency room (A&E)
  * Continence Service consultations (face-to-face visits and/or phone calls)
  * Number of hospital admissions
  * Days spent at hospital
  * Use of relevant medications (including opioids, antidepressants, bladder stabilisers or any other medication inducing constipation) and supplies (diapers, protector sheets, suppositories and micro-enemas) during the 12-week RCT period; and mean/median change in the use of TAI while using Mowoot during the 12-week RCT period
Continence Service consultations (HE outcome) | 3 times during the follow-up: Once at visit 1 (day 14 after recruitment), once at visit 2 (day 42 after treatment), and once more at visit 3 (day 154 after recruitment)
  Quantitative assessment of the changes in the direct medical healthcare costs due to constipation-related problems assessed as the number of continence Service consultations (face-to-face visits and/or phone calls) over the previous 8 weeks
Number of hospital admissions (HE outcome) | 3 times during the follow-up: Once at visit 1 (day 14 after recruitment), once at visit 2 (day 42 after treatment), and once more at visit 3 (day 154 after recruitment)
  Quantitative assessment of the changes in the direct medical healthcare costs due to constipation-related problems assessed as the number of hospital admissions over the previous 8 weeks
Days spent at hospital (HE outcome) | 3 times during the follow-up: Once at visit 1 (day 14 after recruitment), once at visit 2 (day 42 after treatment), and once more at visit 3 (day 154 after recruitment)
  Quantitative assessment of the changes in the direct medical healthcare costs due to constipation-related problems assessed as the days spent at hospital over the previous 8 weeks
Use of relevant medications (HE outcome) | 3 times during the follow-up: Once at visit 1 (day 14 after recruitment), once at visit 2 (day 42 after treatment), and once more at visit 3 (day 154 after recruitment)
  Quantitative assessment of the changes in the direct medical healthcare costs due to constipation-related problems assessed as the use of relevant medications, including opioids, antidepressants, bladder stabilisers or any other medication inducing constipation, over the previous 8 weeks
Use of relevant supplies (HE outcome) | 3 times during the follow-up: Once at visit 1 (day 14 after recruitment), once at visit 2 (day 42 after treatment), and once more at visit 3 (day 154 after recruitment)
  Quantitative assessment of the changes in the direct medical healthcare costs due to constipation-related problems assessed as the use of relevant supplies (diapers, protector sheets, suppositories and micro-enemas), over the previous 8 weeks
Incremental cost/effectiveness ratio (ICER) and Quality-Adjusted Life years (QALYS) (HE outcome) | EQ-5D-5L3 answered 3 times during the follow-up: Once at visit 1 (day 14 after recruitment), once at visit 2 (day 42 after treatment), and once more at visit 3 (day 154 after recruitment)
  Quantitative assessment of the of ICER and QALYS based on the health-related quality of life questionnaire EQ-5D-5L
Adverse events and Serious adverse events | Evrey day during all the follow-up, from recruitment (visit 0, day 0) to the end of study (visit 3, day 154)
  Quantitative and qualitative assessment of adverse events (AEs) and serious adverse events (SAEs)

CONTACTS AND LOCATIONS:
Overall Officials: Immaculada Herrero, PhD, Study Chair — usMIMA S.L.
Locations (3):
- United Kingdom (3):
  - University Hospital of North Durham, NHS Foundation Trust, Durham, County Durham and Darlington
  - University Hospital of North Tees, North Tees & Hartlepool NHS Foundation Trust, Hardwick
  - The Newcastle Upon Tune Hospitals NHS Foundation Trust., Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ayas S, Leblebici B, Sozay S, Bayramoglu M, Niron EA. The effect of abdominal massage on bowel function in patients with spinal cord injury. Am J Phys Med Rehabil. 2006 Dec;85(12):951-5. doi: 10.1097/01.phm.0000247649.00219.c0. PMID 17117000
- [Background] Diego MA, Field T. Moderate pressure massage elicits a parasympathetic nervous system response. Int J Neurosci. 2009;119(5):630-8. doi: 10.1080/00207450802329605. PMID 19283590
- [Background] Sinclair M. The use of abdominal massage to treat chronic constipation. J Bodyw Mov Ther. 2011 Oct;15(4):436-45. doi: 10.1016/j.jbmt.2010.07.007. Epub 2010 Aug 25. PMID 21943617
- [Background] Marquis P, De La Loge C, Dubois D, McDermott A, Chassany O. Development and validation of the Patient Assessment of Constipation Quality of Life questionnaire. Scand J Gastroenterol. 2005 May;40(5):540-51. doi: 10.1080/00365520510012208. PMID 16036506
- [Background] Frank L, Kleinman L, Farup C, Taylor L, Miner P Jr. Psychometric validation of a constipation symptom assessment questionnaire. Scand J Gastroenterol. 1999 Sep;34(9):870-7. doi: 10.1080/003655299750025327. PMID 10522604
- [Background] Drossman DA, Hasler WL. Rome IV-Functional GI Disorders: Disorders of Gut-Brain Interaction. Gastroenterology. 2016 May;150(6):1257-61. doi: 10.1053/j.gastro.2016.03.035. No abstract available. PMID 27147121
- [Background] Yiannakou Y, Tack J, Piessevaux H, Dubois D, Quigley EMM, Ke MY, Da Silva S, Joseph A, Kerstens R. The PAC-SYM questionnaire for chronic constipation: defining the minimal important difference. Aliment Pharmacol Ther. 2017 Dec;46(11-12):1103-1111. doi: 10.1111/apt.14349. Epub 2017 Oct 6. PMID 28983926
- [Background] Forootan M, Bagheri N, Darvishi M. Chronic constipation: A review of literature. Medicine (Baltimore). 2018 May;97(20):e10631. doi: 10.1097/MD.0000000000010631. PMID 29768326
- [Background] Lamas K, Lindholm L, Engstrom B, Jacobsson C. Abdominal massage for people with constipation: a cost utility analysis. J Adv Nurs. 2010 Aug;66(8):1719-29. doi: 10.1111/j.1365-2648.2010.05339.x. Epub 2010 Jun 16. PMID 20557387
- [Background] McClurg D, Booth L, Herrero-Fresneda I. Safety and Efficacy of Intermittent Colonic Exoperistalsis Device to Treat Chronic Constipation: A Prospective Multicentric Clinical Trial. Clin Transl Gastroenterol. 2020 Dec;11(12):e00267. doi: 10.14309/ctg.0000000000000267. PMID 33512794
- [Background] Bremer J, Bremer J, Konig M, Kossmehl P, Kurze I, Obereisenbuchner J, Weinschenk E, Herrero-Fresneda I. Intermittent colonic exoperistalsis for chronic constipation in spinal cord-injured individuals. A long-term structured patient feedback survey to evaluate home care use. Spinal Cord Ser Cases. 2023 Jul 29;9(1):37. doi: 10.1038/s41394-023-00597-z. PMID 37516745
- [Result] Emmanuel A, Kumar G, Christensen P, Mealing S, Storling ZM, Andersen F, Kirshblum S. Long-Term Cost-Effectiveness of Transanal Irrigation in Patients with Neurogenic Bowel Dysfunction. PLoS One. 2016 Aug 24;11(8):e0159394. doi: 10.1371/journal.pone.0159394. eCollection 2016. PMID 27557052